CLINICAL TRIAL: NCT06414239
Title: Amélioration du Taux de succès de la Coloscopie Totale Lors Des Endoscopies Digestives Sans anesthésie : évaluation du Masque de réalité Virtuelle
Brief Title: Improvement of Lower Digestive Endoscopy Without Anesthesia : Evaluation of the Virtual Reality Mask
Acronym: REVENDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP220675
Record Dates: First submitted 2024-04-29; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Digestive System Disease
Keywords: Lower digestive endoscopy whatever the indication; Digestive endoscopy; Colonoscopy; Virtual reality
MeSH Terms: conditions — Digestive System Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Coloscopy with a virtual reality mask
  Interventions: Device: Use of a VR mask
- Control group (Other): Coloscopy without any premedication or anesthesia
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Use of a VR mask — Virtual reality mask
  Arms: Interventional group
Other: Standard of care — Without any premedication or anesthesia
  Arms: Control group

SUMMARY:
90% of colonoscopies are performed with general anesthesia (GA). GA carries risks and requires a prior anesthesia consultation, a dedicated team and technical platform on the day of the examination. These constraints increase the time it takes to organize examinations. This was particularly highlighted during the recent health crisis. The success of colonoscopy without GA varies depending on the patient's experience of the examination. Any measure allowing better tolerance of the exam is therefore likely to increase its success rate and avoid rescheduling the exam under GA. A 2017 meta-analysis showed that the use of virtual reality (VR) reduced pain and anxiety during care for burn victims, in trauma and oncology. In upper digestive endoscopy, retrospective studies have shown good tolerability of the examinations and a reduction in pain compared to patients with only local anesthesia. Thus, if the VR mask improves the success rate of total colonoscopy by improving tolerance and acceptability, more examinations without GA could be considered. It could also have an economic impact.

ELIGIBILITY:
Inclusion Criteria:

Patient over 18 years old with an indication for total colonoscopy and accepting without General Anesthesia

Exclusion Criteria:

* Hearing problems or low vision
* Psychiatric or cognitive disorders hindering communication
* History of epilepsy
* Claustrophobia which can lead to a rejection of the virtual reality mask
* History of cybercynetosis during previous use of VR
* Chronic abdominal pain with baseline Visual analogue scale (VAS) > 5
* Emergency examination
* Patient participating in another interventional research on digestive endoscopy
* Patient not speaking French
* Patient under guardianship

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of cecal intubation | At day 0
  Success of a total colonoscopy defined by the rate of cecal intubation (visualization of the ileocecal valve and the appendicular orifice with the endoscope located near the appendicular orifice) or visualization of the ileocecal anastomosis in case of history of surgery removing the ileocaecal valve

SECONDARY OUTCOMES:
Maximum pain assessed by the patient by numerical scale | At day 0
  The scale varies from 0 to 10. 0 is no pain, 10 is the worst possible pain
Maximum pain assessed by the patient by numerical scale | At 1 month
  The scale varies from 0 to 10. 0 is no pain, 10 is the worst possible pain
Maximum anxiety assessed by the patient by numerical scale | At day 0
  The scale varies from 0 to 10. 0 is no anxiety, 10 is the worst possible anxiety
Maximum anxiety assessed by the patient by numerical scale | At 1 month
  The scale varies from 0 to 10. 0 is no anxiety, 10 is the worst possible anxiety
Patient's opinion to repeat the examination under the same conditions | At day 0
  It will be assesses by the Likert scale
Patient's opinion to repeat the examination under the same conditions | At 1 month
  It will be assesses by the Likert scale
Duration of the examination | At day 0
  Time between introduction and removal of the colonoscope
Total duration of the procedure | At day 0
  time between entering and leaving the room
Number of minutes from visualization of the valve between the introduction of the colonoscope and 30 minutes maximum | At day 0
  Between the introduction of the colonoscope and 30 minutes maximum. It can be the ileum in the event of a history of surgery removing the valve.
Proportion of procedures where the VR mask is removed at the patient's request | Up to 30 months
Proportion of colonoscopies with detection of at least one adenoma | Up to 30 months
Proportion of VR device malfunctions (≥ 1) during the procedure in the intervention group | Up to 30 months
Operator satisfaction | Up to 30 months
  Assessed by the Analogue Visual Scale examination
Incremental cost effectiveness ratio or incremental cost-result ratio in the form of cost per additional colonoscopic success | Up to 30 months